CLINICAL TRIAL: NCT06110741
Title: VaxInnate : Evaluation of the Consequences of Poly Vaccination on Innate Immunity : Applications to a Military Population
Brief Title: Evaluation of the Consequences of Poly Vaccination on Innate Immunity : Applications to a Military Population
Acronym: VaxInnate
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PPRC01; 2023-A01356-39 (Other: IDRCB)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Vaccine Breakthrough Infections
MeSH Terms: conditions — Breakthrough Infections | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample and saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sampling and survey group: This group will complete questionnaires and participate in sample collection.
  Interventions: Other: Blood and saliva sampling; Other: Survey
- Survey group: This group will only complete questionnaires
  Interventions: Other: Survey

INTERVENTIONS:
Other: Blood and saliva sampling — Collecting blood and saliva sample
  Groups: Sampling and survey group
Other: Survey — Collecting data on infectious diseases during the study period

SUMMARY:
In this study, the poly vaccination of military personnel prior to deployment will be analyzed in terms of central, peripheral and long-lasting changes in innate immunity.

Analysis of monocyte immune training induced by vaccination will provide a better understanding of the indirect effects of vaccination and their persistence over time.

ELIGIBILITY:
Inclusion Criteria:

* french military personnel
* >18yo
* overseas deployment scheduled between 30 and 60 days after vaccination session
* adult
* able to give consent

Exclusion Criteria:

* unrectified military personnel
* having received a live vaccine within 6 months prior to inclusion
* having received an attenuated vaccine within 3 months prior to inclusion
* pregnancy or breastfeeding
* vaccine contraindication
* major incapacity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed by healthy subjects which have to receive a vaccine update in order to be deployed
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Monocytes' functional reprogramming | 11 months
  describing the functional reprogramming of monocytes following vaccination sessions among military personnel prior and after deployment

SECONDARY OUTCOMES:
Identify immune signatures | 11 months
  Identifying immune signatures by comparing the functional reprogramming of monocytes by different vaccines and co vaccinations schemes
Time persistence | 11 months
  Assess the persistence over time of the effects by follow-up after return from mission

IPD SHARING:
Plan to Share IPD: No